CLINICAL TRIAL: NCT00629486
Title: Genetic Polymorphisms of Interleukin-1B and TNF-A and HBV-Related Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Fa,Tsai, Professor of Medicine, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KMUH-IRB-950181
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis B; Hepatocellular Carcinoma; Chronic Liver Disease
Keywords: cytokine gene; hepatitis B; hepatocellular carcinoma; chronic liver disease
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular | interventions — Tumor Necrosis Factor-alpha; Polymorphism, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cytokines were determined (Experimental): prevalence of genetic polymorphisms of interleukin 1B was measured in HBV-related hepatocellular carcinoma
  Interventions: Genetic: Polymorphism of IL-1 beta and TNF-alpha

INTERVENTIONS:
Genetic: Polymorphism of IL-1 beta and TNF-alpha — To analyze the role of polymorphisms of IL-1beta and TNF-alpha gene on risk of hepatitis B-related chronic liver disease and hepatocellular carcinoma
  Other Names: polymorphism; TNF-alpha; interleukin-1L

SUMMARY:
By detecting polymorphisms of IL-1β and TNF-α,this study aims to find the effects of cytokine gene polymorphisms(and their interaction) on susceptibility and severity of HBV-related HCC.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV)infection is the major risk factor for chronic liver disease and hepatocellular carcinoma (HCC). Host immunogenetic factors contribute to HBV-associated liver damage and/or carcinogenesis. Variant cytokine alleles, including tumor necrosis factor-α(TNF-α)and interleukin-1β(IL-1β), might contribute to interindividual difference in inflammatory responses and account for heterogeneous disease outcome of infectious disease.

By detecting polymorphisms of IL-1β and TNF-α,this study aims to find the effects of cytokine gene polymorphisms(and their interaction) on susceptibility and severity of HBV-related HCC.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-positive patients

Exclusion Criteria:

* HBsAg-negative patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
cytokine polymorphisms increase risk for hepatocellular carcinoma | years

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Fa Tsai, M.D., Ph.D., Principal Investigator — Professor of Medicine
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Hospital, Kaohsiung City, Kaohsiung
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung